CLINICAL TRIAL: NCT00274742
Title: An Open-label, Multi-center Phase I Study to Investigate the Tolerability and Safety of a Continuous Infusion of the Bispecific T-cell Engager MT103 in Patients With Relapsed Non-Hodgkin's Lymphoma (NHL)
Brief Title: Safety Study of the Bispecific T-cell Engager Blinatumomab (MT103) in Patients With Relapsed NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT103-104
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Non-Hodgkin's Lymphoma, Relapsed
Keywords: Non-Hodgkin's Lymphoma; Cancer immunotherapy; Monoclonal antibody; anti-CD19; anti-CD3; BiTE; Blinatumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Bites and Stings | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): Patients received blinatumomab as continuous intravenous infusion for 4 weeks. Participants with clinical benefit were permitted to continue for another 4 weeks for a total of 8 weeks. Participants with a clinical benefit 4 weeks after completion of the first cycle of treatment could also receive additional treatment approximately 3 months ater the end of infusion at the same dose level.
  Interventions: Biological: Blinatumomab (MT103)

INTERVENTIONS:
Biological: Blinatumomab (MT103) — Doses from 0.5 to 120 µg/m^2/24hours by continuous intravenous infusion
  Other Names: Blinatumomab; MT103; AMG103; BLINCYTO™

SUMMARY:
The purpose of this study is to determine whether a continuous infusion of Blinatumomab (MT103) is safe in the treatment of relapsed Non-Hodgkin's Lymphoma.

Furthermore, the study is intended to provide pharmacokinetic and pharmacodynamic data of Blinatumomab as well as to get first indication of tumour activity.

DETAILED DESCRIPTION:
Non-Hodgkin's Lymphoma (NHL) represents the 6th most common cancer. Globally, around 165,000 new cases are diagnosed each year, with approximately 90,000 deaths per year. The vast majority of NHLs are B-cell derived (90%) and express common B-cell antigens such as CD19, CD20 and CD22. NHL can be divided into indolent (low-grade) and aggressive (high-grade) lymphomas. Still almost all patients with advanced stage indolent disease will die from their disease. Therefore, a high medical need exists to develop novel agents that further improve the survival of NHL patients.

Blinatumomab (MT103) is a bispecific antibody derivative, anti-CD19 x anti-CD3, designed to link B-cells and T-cells resulting in T-cell activation and a cytotoxic T-cell response against CD19+ cells. Data of prior phase I studies show evidence of biological activity in humans. In vitro and ex-vivo data suggest that a longterm presence of the drug in target tissues may provide antitumour activity.

The study investigates the safety and tolerability of different doses of Blinatumomab administration in a continuous infusion regimen. Maximum tolerated dose (MTD) will be defined in a classical 3+3 dose escalation regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first or later relapse of histologically (World Health Organisation classification) confirmed:

   * follicular lymphoma (grade I/II)
   * marginal zone lymphoma
   * lymphoplasmocytic lymphoma
   * mantle cell lymphoma
   * diffuse large B-cell lymphoma
   * small lymphocytic lymphoma requiring therapy and not eligible for curative treatment
2. Measurable disease (at least one lesion >= 1.5 cm) documented by computed tomography (CT) scan
3. Age >= 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status <=2
5. Life expectancy of at least 6 months
6. Ability to understand the patient information and informed consent form
7. Signed and dated written informed consent is available
8. B:T cell ratio (Fluorescence-Activated Cell Sorter [FACS] analysis results by central lab) available before study entry.

Exclusion Criteria:

1. Any other NHL not listed in inclusion criterion 1
2. Abnormal laboratory values as defined below:

   * Peripheral lymphocyte count > 20 x 10^9/L
   * Platelet counts ≤ 75,000/µL
   * Hemoglobin level ≤ 9 g/dL
   * Venous pH value out of normal range or oxygen saturation ≤ 90%
3. Known or suspected central nervous system (CNS) involvement by NHL
4. a)History of or current relevant CNS pathology as epilepsy, seizure, paresis,aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis b)Evidence for presence of inflammatory lesions and/or vasculitis on cerebral MRI
5. Autologous stem cell transplantation within 12 weeks prior to study entry
6. Allogeneic stem cell transplantation
7. Cancer chemotherapy within 4 weeks prior to study entry
8. Radiotherapy within 4 weeks prior to study entry
9. Treatment with rituximab within 4 weeks prior to study entry
10. Prior treatment with alemtuzumab 12 weeks prior to study entry
11. Treatment with any investigational agent within 12 weeks prior to study entry
12. Contraindication for any of the concomitant medications
13. Abnormal renal or hepatic function as defined below:

    * Aspartate aminotransferase (AST; SGOT) and/or alanine aminotransferase (ALT; SGPT) >= 2 x upper limit of normal (ULN)
    * total bilirubin >= 1.5 x ULN
    * serum creatinine >= 2 x ULN
    * creatinine clearance < 50mL/min
14. Indication of hypercoagulative state as defined below:

    -antithrombin activity <LLN
15. Presence of human anti-murine antibodies (HAMA) or known hypersensitivity to immunoglobulins
16. History of malignancy other than B-cell lymphoma within 5 years prior to study entry, with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix
17. Active infection / not yet recovered from recent infection; known bacteriemia
18. Any concurrent disease or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator
19. Regular dose of corticosteroids during the four weeks prior to D1 of this study or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent, or any other immunosuppressive therapy within 4 weeks prior to study entry
20. Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B or hepatitis C virus
21. Pregnant or nursing women, or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least three months thereafter. Male patients not willing to ensure that during the study and at least three months thereafter no fathering takes place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-06; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bargou, MD, PhD, Principal Investigator — Medizinische Poliklinik der Julius-Maximilians-Universität Würzburg, Zentrum für Innere Medizin, Oberdürrbacherstr. 6 D-97080 Würzburg
Locations (5):
- Germany (5):
  - Medizinische Klinik 5, Hämatologie & Internistische Onkologie, Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Klinik für Hämatologie, Medizinische Klinik und Poliklinik, Essen
  - Universtätsklinkum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Abteilung Innere Medizin III, Ulm
  - Medizinische Poliklinik der Julius-Maximilians-Universität Würzburg, Würzburg

REFERENCES:
- [Derived] Nagele V, Zugmaier G, Goebeler ME, Viardot A, Bargou R, Kufer P, Klinger M. Relationship of T- and B-cell kinetics to clinical response in patients with relapsed/refractory non-Hodgkin lymphoma treated with blinatumomab. Exp Hematol. 2021 Aug;100:32-36. doi: 10.1016/j.exphem.2021.06.005. Epub 2021 Jul 3. PMID 34228983
- [Derived] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 22 June 2004 through 18 July 2011
Pre-assignment Details: Participants were enrolled into 20 different cohorts representing different dose levels, modes of administration (ramp, single-step, double-step, flat), or populations. To facilitate the analysis of the study, the different cohorts were grouped into six "dose groups" based on the dose that was intended to be given to a participant.
Groups:
- Blinatumomab ≤ 5 µg/m²/d: Participants received blinatumomab ≤ 5 µg/m²/day as continuous intravenous infusion over 4-8 weeks in the first treatment cycle.
- Blinatumomab 15 µg/m²/d: Participants received blinatumomab 15 µg/m²/day as continuous intravenous infusion over 4-8 weeks in the first treatment cycle.
- Blinatumomab 30 µg/m²/d: Participants received blinatumomab 30 µg/m²/day as continuous intravenous infusion over 4-8 weeks in the first treatment cycle.
- Blinatumomab 60 µg/m²/d Flat: Participants received blinatumomab 60 µg/m²/day without a lower dose as continuous intravenous infusion over 4-8 weeks in the first treatment cycle.
- Blinatumomab 60 µg/m²/d Step: Participants received blinatumomab 60 μg/m²/day as continuous intravenous infusion after initial lower doses of 5 and/or 15 μg/m²/day for a total treatment duration of 4-8 weeks in the first treatment cycle.
- Blinatumomab 90 µg/m²/d: Participants received blinatumomab 90 µg/m²/day as continuous intravenous infusion over 4-8 weeks in the first treatment cycle.
Period: Overall Study
Arm/Group | Blinatumomab ≤ 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d Flat | Blinatumomab 60 µg/m²/d Step | Blinatumomab 90 µg/m²/d
Started | 12 | 13 | 6 | 9 | 32 | 4
Completed | 12 (Participants completed the first treatment and 4-week follow-up.) | 5 (Participants completed the first treatment and 4-week follow-up.) | 4 (Participants completed the first treatment and 4-week follow-up.) | 4 (Participants completed the first treatment and 4-week follow-up.) | 16 (Participants completed the first treatment and 4-week follow-up.) | 1 (Participants completed the first treatment and 4-week follow-up.)
Not Completed | 0 | 8 | 2 | 5 | 16 | 3
Not completed — Adverse Event | 0 | 4 | 1 | 4 | 12 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — End of Study | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 3 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinatumomab ≤ 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d Flat | Blinatumomab 60 µg/m²/d Step | Blinatumomab 90 µg/m²/d | Total
Number analyzed (Participants) | 12 | 13 | 6 | 9 | 32 | 4 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (7.5) | 64.8 (8.0) | 53.3 (9.4) | 59.7 (11.9) | 57.1 (14.9) | 64.8 (5.6) | 60.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 0 | 11 | 1 | 19
  Male | 10 | 9 | 5 | 9 | 21 | 3 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 13 | 6 | 9 | 32 | 4 | 76
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Participants reporting at least one occurence of any adverse event including clinical symptoms, laboratory abnormalities, serious adverse events, and treatment-limiting adverse events
Time Frame: From the first infusion of blinatumomab until the safety follow-up visit 2 weeks after end of the treatment period, including the consolidation and relapse periods. The median treatment duration was 33.24 days.
Population: All participants who received at least one infusion of blinatumomab
Measure: Number; unit: participants
Arm/Group | Blinatumomab ≤ 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d Flat | Blinatumomab 60 µg/m²/d Step | Blinatumomab 90 µg/m²/d
Number analyzed (Participants) | 12 | 13 | 6 | 9 | 32 | 4
participants | 12 | 13 | 6 | 9 | 32 | 4

2. Secondary Outcome: Serum Concentration of Blinatumomab
Description: The steady state serum concentration (Css), summarized as the observed concentrations collected at least 10 hours after the start of continuous intravenous infusion or within the sampling window at the end of infusion. Concentrations below the lower limit of quantitation (100 pg/mL) were excluded from analysis.
Time Frame: Up to 24 hours after the end of infusion.
Population: Participants who received blinatumomab and had available pharmacokinetic data
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Blinatumomab 5 µg/m²/d: Participants who received blinatumomab 5 µg/m²/day as continuous intravenous infusion in the first treatment cycle.
- Blinatumomab 15 µg/m²/d: Participants who received blinatumomab 15 µg/m²/day as continuous intravenous infusion in the first treatment cyle.
- Blinatumomab 30 µg/m²/d: Participants received blinatumomab 30 µg/m²/day as continuous intravenous infusion in hte first treatment cycle.
- Blinatumomab 60 µg/m²/d: Participants received blinatumomab 60 µg/m²/day as continuous intravenous infusion in the first treatment cycle.
- Blinatumomab 90 µg/m²/d: Participants received blinatumomab 90 µg/m²/day as continuous intravenous infusion in the first treatment cycle.
Arm/Group | Blinatumomab 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d | Blinatumomab 90 µg/m²/d
Number analyzed (Participants) | 32 | 36 | 6 | 34 | 4
pg/mL | 210 (84.9) | 651 (307) | 1210 (476) | 2730 (985) | 3490 (904)

3. Secondary Outcome: Objective Tumor Response According to the Cheson Criteria (Without Minimal Response)
Description: Tumor response was defined according to the Cheson criteria and assessed after 4 and 8 weeks of study treatment using computed tomography (CT) scan (neck, thorax and abdomen/pelvic to assess nodal disease/organ enlargement due to nodal/diffuse infiltration), and bone marrow biopsy (to assess bone marrow infiltration).
  Best clinical response is defined as the best response achieved during the course of the study, with response defined as: Complete Response, Complete Response Unconfirmed, Partial Response, Stable Disease, and Progressive Disease. In this analysis minimal response is set to stable disease as intended in the response categories according to the Cheson criteria. An independent external review by a radiologist (computed tomography scans) and a pathologist (biopsies) was performed to confirm response status.
  If no post-baseline tumor assessment was available, the overall clinical response was set to not available.
Time Frame: Assessed after 4 and 8 weeks of treatment
Population: All participants who received at least one infusion of blinatumomab
Measure: Number; unit: participants
Arm/Group | Blinatumomab ≤ 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d Flat | Blinatumomab 60 µg/m²/d Step | Blinatumomab 90 µg/m²/d
Number analyzed (Participants) | 12 | 13 | 6 | 9 | 32 | 4
participants
  Complete response | 0 | 1 | 1 | 3 | 5 | 1
  Complete response unconfirmed | 0 | 0 | 0 | 0 | 5 | 0
  Partial response | 0 | 2 | 0 | 5 | 6 | 1
  Stable disease | 6 | 7 | 2 | 0 | 7 | 1
  Progressive disease | 6 | 3 | 2 | 0 | 7 | 0
  Not available | 0 | 0 | 1 | 1 | 2 | 1

4. Secondary Outcome: Objective Tumor Response According to the Cheson Criteria (With Minimal Response)
Description: Tumor response was defined according to the Cheson criteria and assessed after 4 and 8 weeks of study treatment using computed tomography (CT) scan (neck, thorax and abdomen/pelvic to assess nodal disease/organ enlargement due to nodal/diffuse infiltration), and bone marrow biopsy (to assess bone marrow infiltration). Minimal response was treated as a separate response category in this analysis. Best clinical response was defined as the best response achieved during the course of the study, whereby the following order was applied: Complete Response, Complete Response Unconfirmed, Partial Response, Minimal Response, Stable Disease, and Progressive Disease.
  If no post-baseline tumor assessment was available, the overall clinical response was set to not available.
Time Frame: Assessed after 4 and 8 weeks of treatment
Population: All participants who received at least one infusion of blinatumomab
Measure: Number; unit: participants
Arm/Group | Blinatumomab ≤ 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d Flat | Blinatumomab 60 µg/m²/d Step | Blinatumomab 90 µg/m²/d
Number analyzed (Participants) | 12 | 13 | 6 | 9 | 32 | 4
participants
  Complete response | 0 | 1 | 1 | 3 | 5 | 1
  Complete response unconfirmed | 0 | 0 | 0 | 0 | 5 | 0
  Partial response | 0 | 2 | 0 | 5 | 6 | 1
  Minimal response | 1 | 1 | 1 | 0 | 2 | 1
  Stable disease | 5 | 6 | 1 | 0 | 5 | 0
  Progressive disease | 6 | 3 | 2 | 0 | 7 | 0
  Not available | 0 | 0 | 1 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: From the first infusion of blinatumomab until the safety follow-up visit 2 weeks after end of the treatment period, including the consolidation and relapse periods. The median treatment duration was 33.24 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  Summary of Adverse Events includes only those participants who received at least one dose of investigational product.
Groups:
- Blinatumomab Overall: All participants who received any dose of blinatumomab
Arm/Group | Blinatumomab ≤ 5 µg/m²/d | Blinatumomab 15 µg/m²/d | Blinatumomab 30 µg/m²/d | Blinatumomab 60 µg/m²/d Flat | Blinatumomab 60 µg/m²/d Step | Blinatumomab 90 µg/m²/d | Blinatumomab Overall
Serious Adverse Events (participants affected / at risk) | 8/12 | 10/13 | 6/6 | 9/9 | 22/32 | 4/4 | 59/76
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13 | 6/6 | 9/9 | 32/32 | 4/4 | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab ≤ 5 µg/m²/d (N=12) | Blinatumomab 15 µg/m²/d (N=13) | Blinatumomab 30 µg/m²/d (N=6) | Blinatumomab 60 µg/m²/d Flat (N=9) | Blinatumomab 60 µg/m²/d Step (N=32) | Blinatumomab 90 µg/m²/d (N=4) | Blinatumomab Overall (N=76)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 3 | 0 | 7
Lymphopenia (Blood and lymphatic system disorders) | 3 | 6 | 6 | 7 | 16 | 4 | 42
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 5 | 0 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Apical granuloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 0 | 0 | 4 | 0 | 7
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 4
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2 | 0 | 4
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 2 | 6
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab ≤ 5 µg/m²/d (N=12) | Blinatumomab 15 µg/m²/d (N=13) | Blinatumomab 30 µg/m²/d (N=6) | Blinatumomab 60 µg/m²/d Flat (N=9) | Blinatumomab 60 µg/m²/d Step (N=32) | Blinatumomab 90 µg/m²/d (N=4) | Blinatumomab Overall (N=76)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 2 | 5 | 1 | 16
Basophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 12 | 2 | 17
Leukopenia (Blood and lymphatic system disorders) | 4 | 9 | 2 | 5 | 10 | 2 | 32
Lymphopenia (Blood and lymphatic system disorders) | 6 | 3 | 2 | 7 | 12 | 1 | 31
Monocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 7 | 0 | 9
Neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 2 | 3 | 4 | 1 | 18
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 5 | 4 | 12 | 2 | 27
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 5 | 0 | 7
Eustachian tube disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 4 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 4
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 6 | 0 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 3 | 4 | 5 | 1 | 20
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 5
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 10 | 1 | 17
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 8 | 0 | 14
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 0 | 3 | 1 | 0 | 3 | 0 | 7
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Catheter site pain (General disorders) | 2 | 2 | 1 | 1 | 1 | 0 | 7
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Chills (General disorders) | 1 | 6 | 4 | 4 | 6 | 0 | 21
Face oedema (General disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 5
Fatigue (General disorders) | 4 | 3 | 3 | 3 | 20 | 2 | 35
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 1 | 5 | 5 | 1 | 12
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 5 | 3 | 1 | 2 | 4 | 0 | 15
Pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 2 | 11 | 6 | 9 | 26 | 4 | 58
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 4
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Immunodeficiency (Immune system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Catheter site infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 4
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Genitourinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 2 | 6 | 0 | 12
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1 | 2 | 1 | 2 | 0 | 9
Activated partial thromboplastin time shortened (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 3
Alanine aminotransferase abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 5 | 2 | 1 | 10 | 2 | 25
Antithrombin III decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Aspartate aminotransferase abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 4 | 2 | 2 | 2 | 2 | 16
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Blood amylase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 2 | 5
Blood bilirubin abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 3
Blood calcium decreased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 3
Blood chloride decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 4
Blood fibrinogen decreased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 3
Blood fibrinogen increased (Investigations) | 0 | 1 | 2 | 1 | 5 | 0 | 9
Blood glucose increased (Investigations) | 4 | 2 | 0 | 0 | 1 | 0 | 7
Blood immunoglobulin A decreased (Investigations) | 0 | 4 | 0 | 3 | 9 | 1 | 17
Blood immunoglobulin E decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Blood immunoglobulin G decreased (Investigations) | 0 | 2 | 0 | 1 | 5 | 2 | 10
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood immunoglobulin M decreased (Investigations) | 1 | 2 | 0 | 2 | 5 | 0 | 10
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 1 | 3 | 3 | 1 | 10
Blood potassium decreased (Investigations) | 3 | 0 | 1 | 2 | 8 | 2 | 16
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 3
Blood urea increased (Investigations) | 0 | 2 | 0 | 0 | 2 | 0 | 4
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Blood urine (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 2
C-reactive protein abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 5 | 5 | 5 | 6 | 12 | 3 | 36
Coagulation factor XII level decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 3
Coagulation factor XIII level increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 2 | 4 | 5 | 4 | 2 | 3 | 20
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 4 | 5 | 7 | 1 | 20
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 3
Haemoglobin decreased (Investigations) | 2 | 2 | 0 | 0 | 0 | 0 | 4
Haptoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Immunoglobulins decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Lipase increased (Investigations) | 2 | 2 | 2 | 0 | 2 | 2 | 10
Lymphocyte count decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 3
Mean cell haemoglobin concentration increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Monocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 3
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Protein S decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 2 | 5 | 3 | 10
Protein total increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 3
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Urinary sediment abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 3 | 5 | 2 | 1 | 11 | 3 | 25
Weight increased (Investigations) | 1 | 5 | 4 | 5 | 14 | 3 | 32
White blood cell count decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 3
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 2 | 0 | 7 | 0 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 7 | 16 | 3 | 31
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 2 | 0 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4 | 4 | 0 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 2 | 7 | 0 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 4 | 0 | 0 | 8
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 6 | 1 | 14
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 4 | 0 | 7
Allodynia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 6
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 4
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 3
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 3 | 6 | 0 | 13
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 4 | 4 | 6 | 11 | 3 | 30
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Intention tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 4
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 5 | 7 | 1 | 13
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Communication disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 6
Emotional distress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0 | 4 | 0 | 7
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 5
Haematuria (Renal and urinary disorders) | 1 | 5 | 1 | 4 | 5 | 1 | 17
Proteinuria (Renal and urinary disorders) | 2 | 2 | 1 | 2 | 2 | 0 | 9
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 3 | 3 | 0 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 3 | 0 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 2 | 1 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 11 | 0 | 16
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 2 | 0 | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 6 | 0 | 7
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2 | 2 | 1 | 7
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 6 | 0 | 8
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.